CLINICAL TRIAL: NCT01879917
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Multi-centre Trial of Liraglutide Treatment in Subjects With Newly Diagnosed Type 1 Diabetes.
Brief Title: Liraglutide in Newly Onset Type 1 Diabetes.
Acronym: NewLira
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); Hillerod Hospital, Denmark (Other); Bispebjerg Hospital (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Thomas Dejgaard, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-005317-39; 2012-005317-39 (EudraCT Number); U1111-1137-3221 (Other: WHO)
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: c-peptide; insulin; hypoglycemia; Newly onset; Diabetes; Type 1; Beta cell; Autoimmune; Glucagon; Meal test
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Hypoglycemia; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Active Comparator): 1.8 mg
  Interventions: Drug: Liraglutide
- Saline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo — Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to investigate the effect and safety of liraglutide 1.8 mg once daily compared to placebo for 52 weeks on change in beta-cell function in patients with newly diagnosed type 1 diabetes as an adjunctive therapy to insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes according to WHO criteria diagnosed ≤ 6 weeks before visit 0
* Age 18 - 40 years - both inclusive
* Postprandial C-peptide > 0.2 nmol/l following sustacal meal test
* Able to understand the written patient information and to give informed consent

Exclusion Criteria:

* Type 2 diabetes
* Body mass index <20 kg/m2
* Pregnancy or unwillingness to use safe contraceptives
* Compromised kidney function (eGFR < 60 ml/min/1,73m2), dialysis or kidney transplantation at visit 0
* Liver disease with elevated plasma alanine aminotransferase (ALT) > three times the upper limit of normal at visit 0

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Beta-cell function | 52 weeks
  To investigate the effect and safety of liraglutide 1.8 mg once daily compared to placebo for 52 weeks on change in beta-cell function in patients with newly diagnosed type 1 diabetes as an adjunctive therapy to insulin treatment.

SECONDARY OUTCOMES:
Postprandial glucagon | 52 weeks
  To investigate the effect of liraglutide as compared to placebo for 52 weeks as an adjunctive therapy to insulin treatment on change in Postprandial glucagon levels following sustacal meal test.

OTHER OUTCOMES:
HbA1c | 52 weeks
  To investigate the effect of liraglutide as compared to placebo for 52 weeks as an adjunctive therapy to insulin treatment on change in: HbA1c.
Insulin dose | 52 weeks
  To investigate the effect of liraglutide as compared to placebo for 52 weeks as an adjunctive therapy to insulin treatment on change ininsulin dose.
Weight | 52 weeks
  To investigate the effect of liraglutide as compared to placebo for 52 weeks as an adjunctive therapy to insulin treatment on change in weight.
Remission period | 52 weeks
  To investigate the effect of liraglutide as compared to placebo for 52 weeks as an adjunctive therapy to insulin treatment on change in length of insulin remission period.
Hypoglycemia | 52 weeks
  To investigate the effect of liraglutide as compared to placebo for 52 weeks as an adjunctive therapy to insulin treatment on change in frequency of hypoglycaemic events.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Madsbad, Professor, Study Director — Hvidovre University Hospital
Locations (1):
- Dep. of Endocrinology, Hvidovre University Hospital, Hvidovre, Capital, Denmark